CLINICAL TRIAL: NCT01115998
Title: Learning Early Travel Skills: Effects of Power Mobility on the Development of Young Children With Severe Motor Impairments
Brief Title: Effect of Power Wheelchairs on the Development and Function of Young Children With Severe Physical Disabilities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Irene McEwen, Principal Investigator, University of Oklahoma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07956; USDE #R305T010757 (Other Grant/Funding Number: U.S. Department of Education)
Record Dates: First submitted 2009-03-19; First posted 2010-05-04 (Estimated); Results first posted 2010-05-04 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Cerebral Palsy; Child, Preschool
Keywords: cerebral palsy; wheelchair; disabled children
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Power wheelchair (Experimental)
  Interventions: Other: Power wheelchair
- Control group (Other)
  Interventions: Other: No power wheelchairs

INTERVENTIONS:
Other: Power wheelchair — Children used power wheelchairs for one year. They continued to receive their usual early intervention services.
  Other Names: Invacare Power Tiger wheelchairs
  Arms: Power wheelchair
Other: No power wheelchairs — Children in the control group did not use power wheelchairs. They continued to receive their usual early intervention services.
  Arms: Control group

SUMMARY:
Self-produced locomotion often is limited in children with cerebral palsy and other conditions that cause severe motor impairments. As a result, these children may be at risk for secondary impairments in spatial cognition, communication, social development, and other domains influenced by independent mobility. To compensate, power mobility has increasingly been advocated for young children with severe motor impairments. The study hypotheses were:

1. Children with severe disabilities that prevent independent locomotion who learn to use power mobility devices when they are 14- to 30-months-of-age will have greater communication, social, and cognitive development over a 12-month period, and will demonstrate more competent coping skills than children with the same characteristics who do not use power mobility.
2. Parents of children who use power mobility will view it as a positive influence on their children's lives, and will perceive their children's development to be more mature than the parents of children who do not use power mobility will perceive their children's development.

DETAILED DESCRIPTION:
More extensive description is not desired.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 to 30 months
* Motor impairment that prevents functional independent mobility
* Vision and hearing adequate to use a power mobility device safely.
* Cognitive abilities assessed to be at least equivalent to a 12-month level or alertness and interest in the environment that suggests a trial of power mobility is warranted.

Ages: 14 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2002-06; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene R McEwen, PT, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Mockler SR, McEwen IR, Jones MA. Retrospective Analysis of Predictors of Proficient Power Mobility in Young Children With Severe Motor Impairments. Arch Phys Med Rehabil. 2017 Oct;98(10):2034-2041. doi: 10.1016/j.apmr.2017.05.028. Epub 2017 Jul 5. PMID 28688787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from throughout Oklahoma between February 2002 and December 2003. They were recruited through the statewide early intervention program, parent groups, radio, and contacts with occupational and physical therapists.
Pre-assignment Details: We used a matched pairs design and did not find matches for some of the children before they became too old for the study.
Groups:
- Power Wheelchair: Children were provided custom-fitted Invacare Power Tiger power wheelchairs to use in their homes and communities for 12 months. Parents were primarily responsible for providing practice opportunities and instruction, with the children's early intervention therapists and research staff helping to solve any problems. Parents were asked to: (1) provide the child with daily opportunities to sit in the device with the motor turned on during play; (2) encourage the child to experiment with movement in a relatively large space and not be concerned if the child drove in circles; and (3) avoid telling the child what to do, but rather to let the child ex experiment unless frustrated or unsafe. The importance of parental supervision, as one would supervise any young child, was stressed. The children also received their usual early intervention services, as specified on their individualized family service plans.
- Control Group: The control group did not receive power wheelchairs. They did receive early intervention services as specified on their individualized family service plans.
Period: Overall Study
Arm/Group | Power Wheelchair | Control Group
Started | 17 | 17
Completed | 11 | 11
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Children received usual early intervention services, but no power wheelchair.
- Total: Total of all reporting groups
Arm/Group | Power Wheelchair | Control Group | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 17 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.78 (.45) | 1.85 (.41) | 1.82 (.43)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34.0

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Evaluation of Disability Inventory
Description: Items measure mobility, self-care, and social function using a 2-point scale (0 = unable or limited ability; 1 = capable in most situations). Items measure caregiver assistance on a 6-point scale (0 = total assistance; 5 = independent). We used the change in scaled scores in each area and total scores for analyses. Worst possible scaled score is 0 and the best possible score is 100.
Time Frame: Baseline and 12 months
Population: We did a per protocol analysis for 22 children who completed the study and an intention to treat (ITT) analysis for the 28 children for whom we had complete data at 12 months. The overall results of the ITT analysis did not differ from the per protocol analysis.
Measure: Median (Inter-Quartile Range); unit: Units on scale
Arm/Group | Power Wheelchair | Control Group
Number analyzed (Participants) | 11 | 11
Units on scale
  Mobility functional skills | 14.6 (2.04) [8.6 to 17.1] | 6.4 (3.11) [-2.7 to 15.5]
  Self-care functional skills | 8.0 (0.95) [5.7 to 11.8] | 7.9 (1.68) [1.4 to 8.5]
  Social function functional skills | 4.7 (1.25) [3.3 to 8.4] | 3.0 (1.93) [0 to 8.6]
  Mobility caregiver assistance | 29.2 (2.97) [17.3 to 36.8] | 14.2 (4.00) [1.8 to 28.2]
  Self-care caregiver assistance | 12.3 (3.60) [11.6 to 25.4] | 5.8 (3.45) [0 to 20.7]
  Social function caregiver assistance | 14.8 (3.36) [9.9 to 28.1] | 19.7 (3.96) [0 to 28.1]
Statistical Analysis 1: Comparison: Power Wheelchair vs Control Group; Mobility functional skills Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = 0.02, Wilcoxon Signed-Rank Test — The a priori alpha level was < 0.10 and was not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Power Wheelchair vs Control Group; Self-care functional skills Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = 0.52, Wilcoxon Signed-Rank Test — The a priori alpha level was <0.10 and was not adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Power Wheelchair vs Control Group; Social function functional skills Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = 0.38, Wilcoxon Signed-Rank Test — The a priori alpha level was 0.10 and it was not adjusted for multiple comparisons
Statistical Analysis 4: Comparison: Power Wheelchair vs Control Group; Mobility care giver assistance. Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = 0.03, Wilcoxon Signed-Rank Test — The a priori alpha level was 0.10 and it was not adjusted for multiple comparisons
Statistical Analysis 5: Comparison: Power Wheelchair vs Control Group; Self-care caregiver assistance Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = .006, Wilcoxon Signed-Rank Test; The a priori alpha level was 0.10 and it was not adjusted for multiple comparisons
Statistical Analysis 6: Comparison: Power Wheelchair vs Control Group; Social function caregiver assistance Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = 0.45, Wilcoxon Signed-Rank Test — The a priori alpha level was <0.10 and it was not adjusted for multiple comparisons

2. Primary Outcome: Battelle Developmental Inventory (BDI)
Description: Items measure adaptive, cognitive, communication, motor, and personal-social development using 3-point ordinal scales (0 = does not complete; 1 = partially completes; 2 = completes item). We used change in age equivalent scores for each area and the total scores for analyses. The worst possible scores are 0 months age equivalent and the best possible scores are 95 months age equivalent.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units on scale
Arm/Group | Power Wheelchair | Control Group
Number analyzed (Participants) | 11 | 11
Units on scale
  Adaptive total | 4.0 (1.06) [2.0 to 5.0] | 3.0 (1.05) [0 to 8.0]
  Cognitive total | 4.0 (1.51) [3.0 to 12.0] | 5.0 (0.93) [2.0 to 8.0]
  Communication total | 7.0 (1.53) [0 to 8.0] | 3.0 (0.98) [0 to 7.0]
  Motor total | 2.0 (0.52) [2.0 to 4.0] | 3.0 (0.50) [0 to 3.0]
  Personal-social total | 5.0 (0.93) [4.0 to 9.0] | 6.0 (1.18) [0 to 9.0]
  BDI total score | 6.0 (0.82) [3.0 to 7.0] | 4.0 (0.73) [1.0 to 8.0]
Statistical Analysis 1: Comparison: Power Wheelchair vs Control Group; Adaptive total Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = 0.92, Wilcoxon Signed-Rank Test — The a priori alpha level was <0.10 and it was not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Power Wheelchair vs Control Group; Cognitive total Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = 0.38, Wilcoxon Signed-Rank Test — The a priori alpha level was <0.10 and it was not adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Power Wheelchair vs Control Group; Communication total Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = 0.42, Wilcoxon Signed-Rank Test — The a priori alpha level was <0.10 and it was not adjusted for multiple comparisons
Statistical Analysis 4: Comparison: Power Wheelchair vs Control Group; Motor total Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = 0.57, Wilcoxon Signed-Rank Test — The a priori alpha level was <0.10 and it was not adjusted for multiple comparisons
Statistical Analysis 5: Comparison: Power Wheelchair vs Control Group; Personal-social total Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = 0.69, Wilcoxon Signed-Rank Test — The a priori alpha level was <0.10 and it was not adjusted for multiple comparisons
Statistical Analysis 6: Comparison: Power Wheelchair vs Control Group; BID total score Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p = 0.28, Wilcoxon Signed-Rank Test — The a priori alpha level was <0.10 and it was not adjusted for multiple comparisons

3. Primary Outcome: Early Coping Inventory
Description: We used the reactive and self-initiated behavior scales. We used change in raw scores for analyses. The worst possible raw score for each scale is 16 and the best possible score is 80.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units on scale
Arm/Group | Power Wheelchair | Control Group
Number analyzed (Participants) | 11 | 11
Units on scale
  Reactive Scale | 6.0 [-2.0 to 12.0] | 2.0 [0 to 12.0]
  Self Initiated Scale | 7.0 [2.0 to 16.0] | 7.0 [-1.0 to 12.0]
Statistical Analysis 1: Comparison: Power Wheelchair vs Control Group; Reactive scale Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p > 0.10, Wilcoxon Signed-Rank Test
Statistical Analysis 2: Comparison: Power Wheelchair vs Control Group; Self Initiated Scale Null hypothesis: The change scores of children in the power mobility and control groups will not differ from baseline to 12 months; Test type: Superiority or Other; p > 0.10, Wilcoxon Signed-Rank Test

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Power Wheelchair | Control Group
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Small sample limited power; matched pairs design limited sample size and analyses; not all children were independent using power wheelchair in 1 year; cognitive measure probably unresponsive to changes in children with physical limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes